CLINICAL TRIAL: NCT07331064
Title: A Phase 1 Clinical Trial of Gallium Maltolate for the Treatment of Pediatric Patients With Relapsed or Refractory Pediatric High-Grade Glioma and Atypical Teratoid Rhabdoid Tumor
Brief Title: Gallium Maltolate for the Treatment of Pediatric Patients With Relapsed or Refractory Pediatric High-Grade Glioma and Atypical Teratoid Rhabdoid Tumor
Acronym: GABRIEL
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sarah Rumler (Other)
Responsible Party: Sponsor-Investigator, Sarah Rumler, Principal Investigator, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-Rumler-GABRIEL
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: High Grade Gliomas; Atypical Teratoid Rhabdoid Tumors (ATRT); Diffuse Midline Glioma; DIPG; Diffuse Intrinsic Pontine Gliomas (DIPG)
Keywords: DIPG; HGG; ATRT; DMG; relapse; refractory; progressive; high grade glioma; diffuse midline glioma; diffuse intrinsic pontine glioma; atypical teratoid rhabdoid tumor; brain tumor; pediatric
MeSH Terms: conditions — Recurrence; Glioma; Diffuse Intrinsic Pontine Glioma; Rhabdoid Tumor; Brain Neoplasms | interventions — gallium maltolate

STUDY DESIGN:
Intervention Model Description: a modified 3 + 3 design with 1 + 1 dose escalation where both escalation and de-escalation are possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gallium Maltolate (GaM) Arm (Experimental): single-agent GaM study, single arm.
  Interventions: Drug: Gallium maltolate

INTERVENTIONS:
Drug: Gallium maltolate — oral small-molecule iron mimetic

SUMMARY:
In this study, we want to find out more about the side effects of an investigational drug for relapsed or refractory atypical teratoid rhabdoid tumor and high-grade glioma, Gallium Maltolate (GaM) and what doses of GaM are safe for people to take. Everyone in this study will receive GaM which is still experimental and is not approved by the U.S. Food and Drug Administration. We do not know all the ways that this drug may affect people. We hope the information from this study will help us develop a better treatment for relapsed or refractory atypical teratoid rhabdoid tumor and high-grade glioma in the future.

DETAILED DESCRIPTION:
We hypothesize that Gallium Maltolate (GaM) can be safely administered for the treatment of pediatric patients with pHGGs and ATRTs that have relapsed following primary treatment or are refractory to primary treatment. This, in turn, will be manifested by antineoplastic activity in patients as measured by progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be obtained before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Patients must have a prior histological diagnosis of pediatric high-grade glioma (WHO Grade 3 or 4, including DMG/DIPG) or ATRT (WHO Grade 4) or molecular features of such tumors (per the 6th volume of Central Nervous System Tumors in the 5th edition of the WHO Classification of Tumors).
3. Patients are required to have received standard treatment for their tumor type which is considered to include at least:

   a. pHGG (including DIPG/DMG): maximum safe resection, focal radiotherapy. i. Addition of temozolomide, bevacizumab, or lomustine are considered of standard of care but not a requirement for inclusion.

   ii. Addition of sites of radiotherapy to include all areas of disease as needed are considered standard of care but not a requirement for inclusion.

   b. ATRT: maximum safe resection, radiotherapy (focal or craniospinal), and combination chemotherapy per a nationally-accepted ATRT regimen (such as DFCI-ATRT, COG ACNS0334, or MUV-ATRT).
4. Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately.

   1. Cytotoxic chemotherapy (given systemically or intraventricular/intrathecal) or other anti-cancer agents known to be myelosuppressive ≥21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
   2. Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): ≥7 days after the last dose of agent.
   3. Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade ≤1 (for purposes of this study, bevacizumab is considered an antibody).
   4. Corticosteroids:

   i. If used to modify immune adverse events related to prior therapy, ≥14 days must have elapsed since last dose of corticosteroid.

   ii. If used for symptom management related to tumor edema or elevated ICP, patient should be on a stable dose of corticosteroid for ≥7 days.

   e. Hematopoietic growth factors: ≥14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or ≥ 7 days for short-acting growth factor.

   f. Autologous stem cell infusion, including boost infusion: ≥42 days g. Cellular therapy: ≥42 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells) h. h. Radiation therapy (XRT)/external beam irradiation including protons: ≥14 days after local XRT; ≥30 days after whole brain or craniospinal XRT.
5. Patients must have measurable disease that can be assessed for response to treatment as defined by RAPNO for high-grade gliomas (59), RAPNO for DIPG (60), or RAPNO for medulloblastoma and other leptomeningeal seeding tumors (for ATRT) (61) that incorporates MRI assessment and clinical factors. In the absence of measurable disease, pathologic confirmation of recurrent disease is required (i.e., positive cerebrospinal fluid cytology).
6. Male or female subjects must be 0-17 years of age.
7. Lanksy/Karnofsky performance status ≥50 (refer to Appendix 1). Subjects who are wheelchair-bound because of paralysis will be considered "ambulatory" when they are up in their wheelchair.
8. Patients must have adequate bone marrow function as evidenced by:

   1. An absolute neutrophil count (ANC) of >1,000/µL (stable off any growth factor within one week of study drug administration.
   2. Hemoglobin >8 g/dL.
   3. Platelet count >100,000/µL without transfusion within one week.
9. Patients must have adequate hepatic and renal function based on the following laboratory tests:

   1. ALT ≤ 2 x ULN
   2. AST ≤ 2 x ULN
   3. Alkaline phosphatase ≤ 2 x ULN
   4. Total bilirubin ≤ 2 x ULN
   5. Adequate kidney function (as defined by eGFR >60 mL/min/1.72m2 as calculated by the Bedside Schwartz equation)
10. Patients must be able to swallow liquid (suspension) medication, or have nasogastric or gastric tube present to give medication.
11. Female subjects must meet one of the following:

    1. Premenstrual OR
    2. If subject is of childbearing potential, agree to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21 days after the last dose of study agent, OR
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
12. Male subjects of child-fathering potential must agree to one of the following:

    1. Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
    2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
13. Patients taking oral iron supplements or iron chelators must discontinue these medications at least one week prior to starting GaM since these agents may impact on the efficacy of GaM. Drug-drug interactions between GaM and other concomitant medications have not been reported.

Exclusion Criteria:

1. Presence of other active malignant disease diagnosed within 12 months.
2. Not appropriately recovered from prior therapy as defined by time frames listed in the inclusion criteria (Section 4.5.2.1).
3. Known hypersensitivity to or intolerance to gallium-based medications.
4. Concurrent use of cytotoxic chemotherapy is not permitted.
5. Unstable or severe concurrent medical conditions such as severe heart disease, renal failure, uncontrolled diabetes mellitus, or severe lung disease.
6. History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion.
7. Patients who have not completed all standard-of-care treatments including surgical procedures and radiation therapy.
8. Inability to tolerate an oral medication.
9. Patients who are pregnant or nursing.
10. Patients with any condition which, in the investigator's opinion, makes the patient unsuitable for study participation.

Ages: 0 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2030-11-15 (Estimated); Study Completion 2031-05-15 (Estimated)

PRIMARY OUTCOMES:
GaM tolerance | From start of treatment with GaM to 30 days after completion of treatment with GaM
  Using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 6.0, identify the tolerance of pediatric patients to a specific dose of oral GaM by grading and attribution to GaM of adverse events.
RP2D | From start of treatment with GaM to 30 days after completion of treatment with GaM
  Using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 6.0, define the MTD, recommended phase 2 dose (RP2D), safety and toxicity of oral gallium maltolate.
GaM PK levels | From start of treatment with GaM to 6 months from start of treatment with GaM (for participants who complete 6 months of treatment).
  Measure serum gallium levels at multiple timepoints to calculate pharmacokinetic parameters in pediatric patients

SECONDARY OUTCOMES:
Disease response | Every 8 weeks for the first 8 cycles (i.e. prior to cycles 3, 5, 7) and then every 12 weeks until completion of therapy (i.e. prior to cycles 10, 13, 16, etc) with GaM due to disease progression or removal from study.
  Document radiologic stabilization, improvement, or progression in the size of recurrent or relapsed HGGs and ATRTs as assessed by consensus recommendations from the Response Assessment in Pediatric Neuro-Oncology (RAPNO) for pediatric high-grade gliomas, diffuse intrinsic pontine gliomas, and medulloblastoma and other leptomeningeal seeding tumors.
Survival | From start of treatment with GaM to 12 months from completion of treatment with GaM.
  Document survival times to determine PFS and OS.
Quality of Life Patient Reported Outcomes | From start of treatment with GaM to 12 months from completion of treatment with GaM
  Document quality of life outcomes using validated quality of life measurements for pediatric patients (PROMIS®).

IPD SHARING:
Plan to Share IPD: Yes
measurements of lesions (as obtained from brain/spine magnetic resonance images (MRI), adverse event descriptions and grading (including any laboratory and ancillary testing required to assess safety and health of subjects, such as blood counts, chemistries, liver testing, pulmonary function testing, and electrocardiogram) as defined by CTCAE V5, quality of life questionnaire data, survival times, and PK/biomarker information In regards to PK data, the subjects will have blood samples taken at the following timepoints to measure serum gallium concentration: on day 1 of administration just prior to drug administration, 0.5, 1, 2, 4, 8, and 24 hours post study drug administration. Additional timepoints will include troughs (i.e. just prior to study drug administration for that particular day) on day 15 of cycle 1, and day 1 of each subsequent cycle.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At least annually, or sooner if protocol changes, recruitment details, or amendments change.
Access Criteria: We will not place any restrictions on data and plan to deposit and publish interim results as soon as they are available.
  There may be an embargo on these data depending the journal that accepts our paper with our findings,